CLINICAL TRIAL: NCT02381509
Title: Predicting the Safety and Effectiveness of Inferior Vena Cava Filters
Acronym: PRESERVE
Status: Completed | Type: Observational
Sponsor: Carelon Research (Other)
Collaborators: ALN Implants Chirurgicaux (Unknown); B. Braun Interventional Systems, Inc (Industry); Bard Peripheral Vascular, Inc. (Industry); Cook Group Incorporated (Industry); Cordis US Corp. (Industry); Argon Medical Devices (Industry); Society of Interventional Radiology Foundation (Other); Society for Vascular Surgery (Other)
Responsible Party: Sponsor
Other Study IDs: M01482
Record Dates: First submitted 2015-03-02; First posted 2015-03-06 (Estimated); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: Pulmonary Embolism; Deep Vein Thrombosis
Keywords: inferior vena cava filters
MeSH Terms: conditions — Pulmonary Embolism; Venous Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No

GROUPS / COHORTS (1):
- IVC Filter: IVC filter for the prevention of PE
  Interventions: Device: IVC Filter

INTERVENTIONS:
Device: IVC Filter

SUMMARY:
PRESERVE is a multi-center, prospective, open-label, non-randomized investigation of commercially available IVC filters from 6 manufacturers placed in subjects for the prevention of pulmonary embolism (PE). This study will enroll up to 1,800 IVC filter subjects (with a maximum of 300 subjects per IVC filter brand) at up to 60 sites in the US. The primary objective of this investigational device exemption (IDE) clinical investigation is to evaluate the safety and effectiveness of the commercially available IVC filters (retrievable and permanent) in subjects with clinical need for mechanical prophylaxis of PE with an IVC filter.

DETAILED DESCRIPTION:
The overall goal is to characterize the current practice of IVC filter placement, including the indications, filter type, frequency and success of filter removal, safety of placement initially and in the long term, including filter mechanical stability and caval patency, and the frequency of subsequent episodes of PE and recurrence of DVT. The first steps are to identify the characteristics of use in a broad range of clinical practice settings in the US.

Commercially available IVC filters from 6 manufacturers in the United States will be used. The type of FDA-cleared IVC filter implanted will be left to the discretion of the Principal Investigator at the Site. The following IVC filters will be utilized in this trial:

1. ALN Vena Cava Filter (with and without hook) (ALN Implants Chirurgicaux)
2. Option™ Elite Retrievable Vena Cava Filter (Argon Medical Devices Inc., designed and manufactured by Rex Medical)
3. VenaTech® LP Vena Cava Filter (B Braun Interventional Systems, Inc.) and VenaTech® Convertible™ Vena Cava Filter
4. DENALI® Vena Cava Filter System (DL900F, DL900J) (Bard Peripheral Vascular, Inc.)
5. Cook Günther-Tulip™ Vena Cava Filter (Cook Incorporated)
6. Cordis OPTEASE® Retrievable Vena Cava Filter and Cordis TRAPEASE® Permanent Vena Cava Filter (Cordis Corporation)

Subjects will be evaluated at Procedure, Discharge, 3-months, 6-months (phone), 12-months, 18-months (phone), and 24-months post-procedure. All subjects in whom the IVC filter is removed will be followed for 1-month postretrieval. Mandated follow-up imaging will be performed at 3 months (plain film) and 12 and 24 months (contrast abdominal CT). In addition, clinical visits with physical exam will be performed at 3 months, 12 months and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female, age 18 years or older;
* Requires IVC filter for prevention of pulmonary embolism (PE);
* Provide written informed consent and written HIPAA authorization prior to initiation of study procedures;
* Willing to comply with the specified follow-up

Exclusion Criteria:

* Subject is unable to participate in study evaluations pre- and post-treatment
* Known sensitivity to contrast or serious contrast reaction such as anaphylaxis for which premedication is known to be unsuccessful in alleviating symptoms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects requiring the placement of one of 6 IVC filters for the prevention of PE.
Sampling Method: Non-Probability Sample
Enrollment: 1428 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2020-03-17 (Actual); Study Completion 2021-09-20 (Actual)

PRIMARY OUTCOMES:
Composite safety endpoint of freedom from clinically significant perforation after successful filter placement, filter embolization, caval thrombotic occlusion, deep vein thrombosis, and perioperative serious adverse event | Within first 365 days (± 30 days)
  Clinically significant perforation is defined as protrusion of filter legs through the wall of the IVC causing hemorrhage or hematoma or touching, impressing, or perforating another organ or that triggers the decision to remove the filter; resulting in an attempt to remove the IVC filter or requiring other intervention. Filter embolization is defined as movement of the filter or its components to a distant anatomic site completely out of the target zone after successful filter placement, confirmed by imaging. Caval thrombotic occlusion is defined as presence of an occluding thrombus in the IVC after filter insertion and documented by ultrasound (US), computed tomography (CT), magnetic resonance (MR) imaging, venography, or autopsy; this may be symptomatic or asymptomatic after successful filter placement. Deep vein thrombosis (DVT) is defined as new symptomatic DVT post-deployment, as determined by standard of care imaging. Serious adverse event is defined by ISO 14155.
Composite effectiveness endpoint of procedural and technical success without occurrence of clinically significant pulmonary embolism | At 12-months in-situ or 1-month post-retrieval (whichever comes first)
  New symptomatic PE confirmed by appropriate imaging

SECONDARY OUTCOMES:
Mechanical Stability | At 3-months, 6-months, 12-months, 18-months, 24-months or at the time of filter retrieval
  Defined by absence of: 1) Migration: cephalad movement of the filter >20mm relative to fixed anatomic landmarks compared to the time of placement, 2) Migration: caudal migration of the filter >20mm relative to fixed anatomic landmarks compared to the time of placement, 3) Perforation: >5mm outside apparent cava wall as determined by CT or perforation of adjacent viscera or major vessel, 4) Filter fracture: any loss of a filter's structural integrity (i.e. breakage or separation) documented by imaging or autopsy, 5) Filter embolization: post-deployment movement of the filter or its components to a distant anatomic site completely out of the target zone
Procedure-related complications | At 3-months
  In the judgment of the Principal Investigator
Major adverse events (composite and individual components) | At 3-months, 6-months, 12-months, 18-months, and 24-months
  Defined as death, PE, caval thrombotic occlusion, DVT, clinically significant perforation, retroperitoneal hematoma, or adjacent organ penetration
Filter tilting >15° | At 3-months, 6-months, 12-months, 18-months, 24-months or at the time of filter retrieval
  As determined by appropriate imaging
Filter retrieval | Up to 24-months
  Includes: Attempted retrieval, Successful retrieval, Failed retrieval, Percentage of retrieval success, Complications associated with filter retrieval, Reasons for failed retrieval
Secondary Effectiveness Endpoint for each IVC filter brand tested only if the study is a success (i.e., both primary safety and effectiveness endpoints have been met) | At 12-months
  PE rate

CONTACTS AND LOCATIONS:
Overall Officials: David L. Gillespie, MD, FACS, Study Chair — Cape Cod Hospital; Matt Johnson, MD, Study Chair — Indiana University School of Medicine
Locations (53):
- United States (53):
  - University of Arkansas, Little Rock, Arkansas
  - Ronald Regan UCLA Medical Center, Los Angeles, California
  - Palo Alto VA, Palo Alto, California
  - University of California San Francisco, San Francisco, California
  - Harbor-UCLA Medical Center, Torrance, California
  - University of Colorado, Aurora, Colorado
  - Yale New Haven Hospital, New Haven, Connecticut
  - Medstar Georgetown, Washington D.C., District of Columbia
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - The Heart Institute Largo, Largo, Florida
  - University of Miami Hospital and Clinics/Jackson Memorial, Miami, Florida
  - Florida Hospital, Orlando, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Tallahasse Memorial Hospital, Tallahassee, Florida
  - St. Mary's Medical Center, West Palm Beach, Florida
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Carle Heart & Vascular Institute, Urbana, Illinois
  - Indiana University, Indianapolis, Indiana
  - LSU Health Sciences Center at Shreveport, Shreveport, Louisiana
  - Boston Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Southcoast Hospital, North Dartmouth, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - St. Louis University, St Louis, Missouri
  - Washington University, St Louis, Missouri
  - Hackensack UMC, Hackensack, New Jersey
  - Overlook Medical Center, Summit, New Jersey
  - Albany Medical Center, Albany, New York
  - Feinstein Institute, Manhasset, New York
  - Mount Sinai Hospital, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - NY Presbyterian Weil Cornell Medical Ctr, New York, New York
  - Rochester Regional Health System, Rochester, New York
  - University Hospital/SUNY Upstate, Syracuse, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Duke Medical Center, Durham, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Miami Valley Hospital/Wright State University, Dayton, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - University of Oklahoma-Tulsa, Tulsa, Oklahoma
  - Oregon Health & Science Center, Portland, Oregon
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Rhode Island Hospital/Miriam Hospital, Providence, Rhode Island
  - Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - UT Southwestern, Dallas, Texas
  - Memorial Hermann Hospital, Houston, Texas
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Medical College of WI/Froedtert Memorial Lutheran Hospital, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Johnson MS, Spies JB, Scott KT, Kato BS, Mu X, Rectenwald JE, White RA, Lewandowski RJ, Khaja MS, Zuckerman DA, Casciani T, Gillespie DL. Predicting the Safety and Effectiveness of Inferior Vena Cava Filters (PRESERVE): Outcomes at 12 months. J Vasc Surg Venous Lymphat Disord. 2023 May;11(3):573-585.e6. doi: 10.1016/j.jvsv.2022.11.002. Epub 2023 Feb 23. PMID 36872169
- [Derived] Johnson MS, Spies JB, Scott KT, Kato BS, Mu X, Rectenwald JE, White RA, Lewandowski RJ, Khaja MS, Zuckerman DA, Casciani T, Gillespie DL. Predicting the Safety and Effectiveness of Inferior Vena Cava Filters (PRESERVE): Outcomes at 12 months. J Vasc Interv Radiol. 2023 Apr;34(4):517-528.e6. doi: 10.1016/j.jvir.2022.12.009. Epub 2023 Feb 23. PMID 36841633